CLINICAL TRIAL: NCT02541838
Title: High Intensity Muscle Power and Balance Perturbation Training to Enhance Balance and Mobility in People With Type 2 Diabetic Peripheral Neuropathy
Brief Title: Enhance Balance and Mobility in People With Type 2 Diabetic Peripheral Neuropathy
Acronym: DPN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: VA Maryland Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Odessa Addison, DPT, PhD, Associate Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00064233
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Complications; Diabetic Neuropathies
Keywords: Autonomic Neuropathy; diabetes; balance control
MeSH Terms: conditions — Diabetes Complications; Diabetic Neuropathies; Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Muscle, Balance, and aerobic exercise (Experimental): This trial will have a single experimental arm that will include the following interventions: Leg muscle strengthening, balance training using balance perturbations, and aerobic exercise. All individuals in this trial will receive all interventions listed.
  Interventions: Other: Muscle power; Other: balance perturbation; Other: aerobic exercise

INTERVENTIONS:
Other: Muscle power
Other: balance perturbation
Other: aerobic exercise

SUMMARY:
Type 2 diabetes results in a host of neuromuscular, muscular, and autonomic system impairments that accelerate age-associated limitations in functional independence and the risk of falls. Diabetic peripheral neuropathy (DPN) contributes to functional declines in balance and mobility because of limitations metabolic abnormalities. The constellation of impairments accompanying type 2 diabetes diminishes muscle function and performance including strength and power. Loss of strength at higher speeds of movement (deficit in power) occurs in neural activation of muscles, changes in muscle properties, and through in older individuals with DPN compared to older controls. Consequently, this deficit in speed dependent muscle power production leads to limitations in rapidly responding to sudden loss of balance stability to prevent falling. The goal of this pilot research program is to determine the feasibility and effectiveness of a mechanism-based therapeutic intervention fro improving balance and mobility functions and preventing falls in older adults with DPN. The investigators pan to use the results from this pilot study to design and implement a larger randomized control trial.

DETAILED DESCRIPTION:
The long-term goal of this research is to establish the effectiveness of a mechanism-based therapeutic intervention for improving balance and mobility functions and preventing falls in older adults with type 2 diabetic peripheral neuropathy (DPN).

Specific Aim 1 will determine if combined high intensity isolated leg muscle power exercise with balance perturbation training (ActiveStep) and aerobic exercise achieves greater improvements in balance stabilization (protective stepping behavior and kinematics) and mobility function (gait parameters and timed functional measures) than a lifestyle based intervention that primarily focuses on aerobic exercise through underlying mechanisms of improved neuromuscular activation (rate and magnitude) and sensorimotor control, improved muscle quality, and increased blood flow to enhance neuromuscular and sensorimotor performance in people with DPN.

Specific Aim #2: To determine if a neuromotor balance training program combined with muscle power exercise training and aerobic exercise, leading to improved neuromuscular and sensorimotor mechanisms, is more effective in improving clinical tests of balance and mobility functions in those with DPN compared with a traditional exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* HbA1C of 5.7% to 9.0% or a fasting blood glucose of greater than or equal to 100
* Participants that are diabetic should be stable on medications for at least 3 months prior to entering the study
* Neuropathy is most likely caused by impaired glucose regulation determined by medical or family history
* Autonomic neuropathy as defined by Toronto Neuropathy Expert Group 2010/2011 consensus criteria
* Medically stable at time of enrollment as determined by screening process

Exclusion Criteria:

* Neuropathy due to factors other than impaired glucose regulation determined by screening process
* Other severe medical illness or condition that would preclude safe participation in the study as determined by the study team
* Severe Autonomic Neuropathy that would limit study participation
* Musculoskeletal limitations that would preclude participation in balance assessment of protective stepping

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Muscle size as determined with a CT Scan from baseline to 3 months and baseline to 6 months | baseline, 3 months, and 6 months
  A Computed Tomography Scan will be used to measure the cross sectional area of the leg muscles in cm. Changes from baseline to 3 and 6 months will be examined.
Change in leg muscle strength as determined with a physiological test from baseline to 3 months and baseline to 6 months | baseline, 3 months, and 6 months
  A strength testing machine will be used to test the strength of the legs in newton meters. Changes from baseline to 3 and 6 months will be examined.
Change in cardiac autonomic neuropathy as determined by heart rate variability from baseline to 3 months and baseline to 6 months | baseline, 3 months, and 6 months
  heart rate variability will be measured by placing electrodes near the heart similar to an EKG. Changes in heart rate variability from baseline to 3 and 6 months will be examined.
Change in protective stepping as determined by the number of steps it take to recover from a balance perturbation from baseline to 3 months and baseline to 6 months | baseline, 3 months, and 6 months
  A machine that pulls individuals side to side will be used to measure the number of steps required to recover balance after a pull. Changes from baseline to 3 and 6 months will be examined.

SECONDARY OUTCOMES:
Change in clinical balance as measured by the Four Square Step Test | baseline, 3 months, and 6 months
  The Four Square Step Test (FSST) will be used to evaluate changes in clinical balance. The FSST is a single item, evaluator-administered tool that assesses the ability to change directions while stepping. It requires the individuals to move in the anterior-posterior and medial-lateral directions while stepping. Changes from baseline to 3 and 6 months will be examined.
Change in mobility as measured by the modified physical performance test | baseline, 3 months, and 6 months
  The modified physical performance test will be used to evaluate changes in mobility. This test requires individuals to perform a variety of every day tests such as going up and down the stairs, standing from a chair, and putting on a coat. Changes from baseline to 3 and 6 months will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Odessa Addison, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of Maryland School of Medicine, Baltimore, Maryland
  - VA Maryland Health Care System, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No